CLINICAL TRIAL: NCT06374550
Title: Jump Start on the Go: Improving Resiliency and the Social-Emotional Development of At-Risk Preschool Children in Childcare Centers Using a Mobile Application
Brief Title: Jump Start on the Go: Improving Resiliency and the Social-Emotional Development of At-Risk Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ruby Natale, Associate Professor of Clinical Pediatrics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20231026
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jump Start on the Go Group (Experimental): Participants will be in this group for a total of up to 12 months. These participants will receive the intervention via a mobile app.
  Interventions: Behavioral: Jump Start on the Go
- Jump Start plus Coronavirus Support Group (Active Comparator): Participants will be in this group for a total of up to 12 months.
  Interventions: Behavioral: Jump Start Plus Coronavirus Support

INTERVENTIONS:
Behavioral: Jump Start on the Go — Centers will receive the Jump Start On The Go mental health program via a mobile app. This will entail receiving 12-24 mental health consultation sessions in which a licensed mental health consultant will use a mobile app that will provide directors and teachers with access to information such as videos, infographics, and an Artificial Intelligence Chatbot on how to work with children with challenging behaviors. Participants will receive the intervention once per week for up to 1 hour.
  Arms: Jump Start on the Go Group
Behavioral: Jump Start Plus Coronavirus Support — The Jump Start Plus Coronavirus Support intervention is a resiliency program that provides behavior management and safety programs administered weekly via zoom.
  Arms: Jump Start plus Coronavirus Support Group

SUMMARY:
The purpose of this study is to test the Jump Start on the Go (JS Go), an app-based program and see how helpful it is at improving resiliency and behavior support within childcare settings.

ELIGIBILITY:
Centers Inclusion Criteria:

1. Centers must have >30 children ages 2-to-5
2. Center must serve low income families
3. Centers must reflect the ethnic diversity of the Miami Dade County Public School System (60% Hispanic, 20% Non-Hispanic Black, 20% Non-Hispanic White).

Participants Inclusion Criteria:

1. Participants must speak English or Spanish or Creole
2. Parents must have a child enrolled in the childcare center that is participating in the study.
3. Children ages 2-5: Parent reported data (name, Date of Birth, behaviors)

Exclusion Criteria:

1. any participants who do not speak English or Spanish or Creole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in classroom practices as measured by Health Environment Rating Scale | Baseline, 2 months after baseline, and up to 1 year
  The Health Environment Rating Scale is a measure with a range of score from 0 to 70 with higher score indicating better classroom practices.

SECONDARY OUTCOMES:
Change in child behaviors as measured by Devereux Early Childhood Assessments (DECA) | Baseline, 2 months after baseline, and up to 1 year
  The Devereux Early Childhood Assessments is a measure with a range of score from 0 to 100 with higher score on Behavior Concerns indicating more problem behaviors.
Change in child behaviors as measured by Strengths and Difficulties Questionnaire (SDQ) | Baseline and up to 1 year
  The Strengths and Difficulties Questionnaire is a total difficulties score that ranges from 0 to 40 with higher scores indicating less child behavior concerns.
Change in resiliency as measured by Brief Resiliency Coping Scale | Baseline and up to 1 year
  The Brief Resiliency Coping Scale is a total score that ranges from 4 to 20 with higher scores indicating higher levels of coping
Change in stress as measured by Childcare Worker Job Stress Index | Baseline and up to 1 year
  The Childcare Worker Job Stress Index is a total score that ranges from 22 to 110 with higher scores indicating higher levels of stress
Change in stress as measured by Everyday Stressors Index | Baseline and up to 1 year
  The Everyday Stressors Index is a total score that ranges from 0 to 80 with higher scores indicating higher levels of stress.
Change in satisfaction as measured by Teacher Opinion and Satisfaction survey | Baseline and up to 1 year
  The Teacher Opinion survey is a measure with a range of score from 12 to 44 with higher score indicating better self-efficacy as it relates to teaching practices.
Mobile Application satisfaction as measured by the Mobile Application Rating Scale | 2 months after baseline
  The Mobile Application Rating Scale is a measure with a range of scores from 29-145 with higher score indicating better engagement, functionality, aesthetics, and information quality, as well as application subjective quality.

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Natale, PhD, PsyD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No